CLINICAL TRIAL: NCT02279459
Title: Dual-Energy CT in Patients With Head and Neck Squamous Cell Carcinomas: Assessing Tumor Perfusion and Prediction of Treatment Outcomes
Brief Title: Dual-Energy CT in Patients With Head and Neck Squamous Cell Carcinomas
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140728-01H
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patients head and neck CT scans performed as standard of care done prior to radiation treatment and approximately 12 weeks following treatment, will be acquired in the dual-energy computed tomography (DECT) mode. Participants will have one additional scan, also in the DECT mode, 2 to 3 weeks after the start of their radiation treatment.

SUMMARY:
The purpose of this study is to utilize dual-energy computed tomography (DECT) to investigate changes in tumor iodine concentration in patients with head and neck squamous cell carcinomas (HNSCC). Dual-energy computerized tomography could easily replace a standard CT neck with the added benefit of providing functional information that would only be possible with advanced computerized tomography perfusion, magnetic resonance diffusion (MRI) or positron emission tomography (PET) imaging techniques.

DETAILED DESCRIPTION:
Patients with head and/or neck tumors routinely have head and neck imaging completed with a computerized tomography scan, commonly called a CT scan. A CT scan combines a series of x-ray views that are taken from many different angles and uses computer processing to create cross-sectional images inside your body. These cross-sectional images are very thin slices, often less than 1 mm thick and allow the radiologist to examine parts of your tissue very closely.

Dual energy computed tomography (DECT) is a fairly new technology that uses both the normal x-ray and also a second less powerful x-ray to make the images. The Ottawa Hospital has scanners in use that are able to take the images that oncologists typically order for patients and can also be set to obtain DECT images at the same time.

The purpose of this study is to investigate whether DECT images can provide helpful information to better predict how the tumor will respond to treatment and the likely course of head and neck tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* untreated, histologically confirmed head and neck squamous cell carcinoma

Exclusion Criteria:

* paranasal sinus involvement of head and neck squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged 18 years and older with untreated, histologically confirmed head and neck squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Correlate iodine quantification with the microvascular density in the biopsy specimen | up to 18 months

SECONDARY OUTCOMES:
Utility of dual-energy computerized tomography obtained during chemoradiation therapy to predict treatment response. | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Santanu Chakraborty, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada